CLINICAL TRIAL: NCT05477498
Title: Iron Substitution With Ferric Carboxymaltose as Treatment Strategy for Heart Failure Patients With Preserved Ejection Fraction: A Prospective, Double-blind, Randomized, Placebo-controlled Trial
Brief Title: Iron Substitution With Ferric Carboxymaltose as Treatment Strategy for Heart Failure Patients With Preserved Ejection Fraction
Acronym: IRON-HFpEF
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Principal Investigator left institution
Sponsor: Cantonal Hosptal, Baselland (Other)
Collaborators: Clinical Trial Unit, University Hospital Basel, Switzerland (Other)
Responsible Party: Principal Investigator, Maria Bösing, Principal Investigator, Cantonal Hosptal, Baselland
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2018-02280
Record Dates: First submitted 2019-07-05; First posted 2022-07-28 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Heart Failure With Normal Ejection Fraction; Iron-deficiency
Keywords: Exercise tolerance; iron substitution
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — ferric carboxymaltose; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Intervention group: Active treatment with ferric carboxymaltose, given as diluted solution by intravenous injection Control group: Placebo, administered as normal saline 0.9%
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Each administration of the study drug will be carried out after completion of all applicable study related assessments. FCM is a dark brown solution and cannot be easily masked from placebo (0.9% saline). Therefore, unblinded study personnel (at least one study nurse) who will not be involved in any study procedures for efficacy or safety will be responsible for preparing the infusion and packing bag and tube in an opaque wrapping. Preparation and wrapping will take place in a different room to maintain subject blinding. Administration of the study drug will take place by blinded study personnel. The results of the central laboratory on iron deficiency status and Hb will be sent only to the unblinded study personnel, who will be responsible for evaluating these parameters for subsequent dosing and/or other intervention, if applicable.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Iron substitution (Experimental): Iron deficiency status will be assessed at the baseline visit (Day 0) as well as after 6 weeks of iron substitution (Week 6). The study drug will be given as FCM solution (Ferinject®, Vifor Pharma AG, Villars-sur-Glâne, Switzerland) by intravenous injection. Infusions of 10 or 20 mL (which is the amount of FCM that is equivalent to 500 or 1000 mg of iron, respectively) will be administered in ≥6 minutes diluted in ≈100 mL of sterile 0.9% sodium chloride solution (NaCl) for 10 mL, or in ≥15 minutes diluted in ≈200 mL for 20 mL. Dosing will be based on screening Hb level and weight, rather than on ferritin and TSAT results. On Day 0 (baseline visit), patients with Hb ≤14 g/dL, both <70 kg and >70 kg will receive 1000 mg FCM (20 mL), whereas patients with Hb >14g/dL will receive 500 mg FCM (10 mL).
  Interventions: Drug: Ferric carboxymaltose
- Placebo (Placebo Comparator): Patients in the control group will receive a placebo solution administered as normal saline (0.9% weight/volume (w/v) NaCl) by intravenous injection as per the instructions for active treatment.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ferric carboxymaltose — Application of FCM solution (Ferinject®, Vifor Pharma AG, Villars-sur-Glâne, Switzerland) by intravenous injection.
  Other Names: Ferinject®
  Arms: Iron substitution
Drug: Placebo — Application of placebo solution administered as normal saline (0.9% weight/volume (w/v) NaCl) by intravenous injection as per the instructions for active treatment.
  Other Names: NaCl 0.9%
  Arms: Placebo

SUMMARY:
This study aims to investigate the effects of treatment with intravenous ferric carboxymaltose on exercise tolerance measured as VO2peak in patients with HFpEF and iron deficiency, compared to placebo.

DETAILED DESCRIPTION:
Iron deficiency is a common comorbidity associated with chronic heart failure (HF) in both, patients with preserved (HFpEF) and reduced ejection fraction (HFrEF), which has unfavorable clinical and prognostic effects. Previous studies have confirmed that HF patients with iron deficiency have a lower exercise tolerance than those without iron deficiency. In iron deficient patients with HFrEF, treatment with intravenous ferric carboxymaltose (FCM) improved symptoms, exercise tolerance and quality of life (QoL). Since the latest guidelines published by the European Society of Cardiology (ESC) in 2016, iron substitution is an official class IIa recommendation in HFrEF, while it has not yet been endorsed in the treatment guidelines for HFpEF. To date, no evidence is available on iron supplementation in HFpEF. Therefore, a clear rationale exists for examining the effects of correcting iron deficiency in this high-risk and steadily growing patient group.

The proposed study will be a single-centre, prospective, double-blind, randomized, placebo-controlled trial in a primary care setting including 86 patients with stable HFpEF and iron deficiency. Participants will undergo three study visits: a baseline visit, a status control visit, and a post-intervention visit. At the baseline visit, measurements of exercise tolerance (using spiroergometry), laboratory parameters and disease-specific biomarkers (using blood samples), tHb-mass (using the carbon monoxide rebreathing method), cardiac and arterial vessel structure and function (using electrocardiogram, echocardiography and PVW), QoL (using 3 validated questionnaires), body composition (using BMI and WHR), and habitual physical activity (using a wrist-worn accelerometer) will be performed. Then, patients randomized to the treatment group will receive FCM (Vifor Pharma AG, Villars-sur-Glâne, Switzerland), whereas those in the control group will receive placebo. At week 6, iron deficiency status will be re-evaluated in all patients and, if necessary, another application of FCM or placebo will be administered, respectively. After the 12-week treatment period, the study measurements will be repeated in all patients (post-intervention visit) to investigate the effects of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent as documented by signature
* NYHA functional classes II-III
* Signs and symptoms of chronic HF, such as:
* Dyspnea
* Paroxysmal nocturnal dyspnea
* Reduced exercise tolerance
* Fatigue
* Extended recovery after exercising
* Peripheral edema (lower leg, ankle)
* EF (ejection fraction) >50%
* Structural or functional changes in echocardiography:
* Left atrial volume index (LAVI) >34 ml/m2 OR
* Left ventricular mass index (LVMI) >115 g/m2 (men), >95 g/m2 (women) OR
* E/E' (ratio between mitral peak velocity of early filling (E) to early diastolic mitral annular velocity (E')) >13 AND mean E' septal and lateral wall <9 cm/s
* NT-proBNP >125 pg/ml
* At least 4 weeks on stable medical treatment or without signs and symptoms of cardiac decompensation
* Iron deficiency defined as:
* Ferritin <100 ng/ml OR
* Ferritin <300 ng/ml with a transferrin saturation (TSAT) <20%

Exclusion Criteria:

* Age <18 years
* Pregnancy or lactation
* Life-expectancy <6 months
* Planned cardiac interventions in the following 6 months
* Unstable angina pectoris
* Uncontrolled brady- or tachyarrhythmia
* Severe uncorrected valvular heart disease
* Paroxysmal atrial fibrillation
* Clinically significant concomitant disease states (e.g. hypertension grades 2-3 (>160/100 mmHg), severe renal failure (GFR <30 ml/min/1.73m2), hepatic dysfunction (ALT or AST >3x upper limit of normal, chronic obstructive pulmonary disease (COPD) grades III-IV)
* On-going cancer treatment
* Significant musculoskeletal disease limiting exercise tolerance
* Active infection
* Immunosuppressive medical therapy
* Earlier hypersensitivity to parenteral iron preparation
* Anemia and iron deficiency due to active and/or chronic bleeding
* Blood transfusion within the previous 30 days
* Red cell, folate and vitamin B12 deficiency
* Known or suspected non-compliance, drug or alcohol abuse
* Inability to follow the procedures of the study, e.g. due to insufficient language skills, psychological disorders, dementia, etc.
* Participation in another intervention study
* Enrolment of the investigators, their family members, and other persons involved in the study procedures
* Hemoglobin < 120 ng/ml in male patients or < 110 ng/ml in female patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2022-08-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in peak oxygen uptake (VO2peak) | 12 weeks
  Change of VO2peak will be measured by spiroergometry at the baseline and post-intervention visit.

SECONDARY OUTCOMES:
Change in ventriculo-arterial coupling (VAC) | 12 weeks
  VAC is defined as the ratio of arterial elastance (Ea) and end-systolic elastance (Ees) and will be approximated echocardiographically based on the method described by Antonini-Canterin et al.
Change in arteriovenous oxygen difference (Da-vO2) | 12 weeks
  Da-vO2 will be calculated using the Fick Principle
Change in pulse wave velocity (PWV) | 12 weeks
  PWV will be measured at the same time as the echocardiographic parameters with the VaSera VS-2000 Vascular Screening System (Fukuda Denshi Co. Ltd, Tokyo, Japan) and evaluated by experienced blinded members of the study team.
Change in New York Heart Association (NYHA) functional class | 12 weeks
  NYHA functional class will be determined according to the New York Heart Association classification.
Change in habitual physical activity | 12 weeks
  Habitual physical activity will be measured by an accelerometer over a period of 14 consecutive days for 24 hours per day following baseline and post-intervention visits. Patients will wear a waterproof micro-electromechanical triaxial activity bracelet on the non-dominant wrist (GeneActiv, Activinsights Ltd, Kimbolton, Cambridgeshire, UK) to assess physical activity intensity (light, moderate, vigorous) and periods of inactivity, sleep and wake.
Change in body composition measured by body mass index (BMI) | 12 weeks
  BMI will be calculated from measured height in meters and weight in kilograms. Weight and height will be combined to report BMI in kg/m^2.
Change in baseline body composition measured by waist to hip ratio (WHR) | 12 weeks
  WHR will be calculated from measured waist circumference (WC) and hip circumference (HC) in centimetres. WC will be divided by HC to report WHR.
Change in total hemoglobin mass (tHb-mass) | 12 weeks
  tHB-mass will be measured with the carbon monoxide (CO)-rebreathing method
Change in quality of life (QoL) by the 36-Item Short Form Health Survey (SF-36) | 12 weeks
  The SF-36 consists of 36 items, which are formatted as binary questions or as semantic 6-point differential scales. It refers to the past 4 weeks and includes 9 content areas concerning vitality, general health perception, physical functioning, social functioning, role limitations (emotional/physical problems), pain, mental health and health change.
Change in baseline quality of life (QoL) by the Kansas City Cardiomyopathy Questionnaire (KCCQ) at 12 weeks. | 12 weeks
  The KCCQ consists of 15 items concerning overall symptoms, emotional, social and mental status within the past 2 weeks.
Change in quality of life (QoL) by the Minnesota Living with Heart Failure Questionnaire (MLWHFQ) at 12 weeks. | 12 weeks
  The MLWHFQ refers to the past 4 weeks and includes 21 questions on a 6-point scale with a maximum of 105 points (<24 good QoL, >45 poor QoL).

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Dieterle, MD, Principal Investigator — University Department of Internal Medicine, Cantonal Hospital Baselland

IPD SHARING:
Plan to Share IPD: Yes
Patient-level anonymised datasets can be requested after completion of all planned analyses and publications from the study centre (anticipated by mid 2022). Public access to the study protocol will be granted by publishing it in a scientific journal.